CLINICAL TRIAL: NCT01831635
Title: Myeloproliferative Neoplasms: an In-depth Case-control Study
Acronym: MOSAICC
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); University of Manchester (Other); Western Australian Institute for Medical Research (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dr Lesley Anderson, Chief Investigator, Queen's University, Belfast
Other Study IDs: B12/24; MPDVOICE001 (Other Grant/Funding Number: MPD Voice)
Record Dates: First submitted 2013-03-27; First posted 2013-04-15 (Estimated); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis
Keywords: case-control; recruitment; response rates; incentives
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Venous blood sample (up to 12 ml) - whole blood, DNA Saliva (2ml) Dried Blood spots (500 µl) Toe-nails (2 great toe-nail clippings)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Myeloproliferative neoplasm case: Patients with Polycythemia vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF) will be recruited based on the WHO diagnostic criteria.
  Exclusion Criteria
  * younger than 18 years old.
  * where the clinician/General Practitioner (GP) does not provide consent.
  * incapable of giving informed consent.
  * physically or cognitively incapable of completing the questionnaire.
  * too ill to participate.
  We will assess whether a pen (branded, non-branded or none), a £10 cheque and/or a charity branded trolley token will affect uptake rates in the study.
  Interventions: Other: Methodological pens; Other: Methodological compensation; Other: Methodological trolley tokens
- General Practice Control: GP controls will be randomly selected and frequency matched to the distribution of cases by 5-year age band, geographic location (Belfast and Southampton) and gender.
  The following patient groups will be excluded. Those:
  * younger than 18 years old.
  * where the clinician/GP does not provide consent.
  * incapable of giving informed consent.
  * physically or cognitively incapable of completing the questionnaire.
  * too ill to participate.
  We will assess whether a pen (branded, non-branded or none), a £10 cheque (at study completion) and/or a charity branded trolley token will affect uptake rates in the study.
  Interventions: Other: Methodological pens; Other: Methodological compensation; Other: Methodological trolley tokens
- Non-blood relative or family Control: Recruitment of 100 non-blood relative/friend controls will be undertaken by asking cases to pass on a flyer to up to 2 or 3 non-blood relatives/friends aged 18 years or older.
  We will assess whether a pen (branded, non-branded or none) and/or a £10 cheque (at study completion) will affect uptake rates in the study. Only a limited number of trolley tokens were available so not assessed in this group.
  Interventions: Other: Methodological pens; Other: Methodological compensation

INTERVENTIONS:
Other: Methodological pens — Randomisation of branded pen, non-branded pen and no pen
Other: Methodological compensation — Randomisation of a £10 monetary reimbursement for expenses on completion of the study
Other: Methodological trolley tokens — Trolley tokens to be randomly assigned to half of cases and General Practice controls.
  Groups: General Practice Control; Myeloproliferative neoplasm case

SUMMARY:
There is a paucity of data on the aetiology of myeloproliferative neoplasms (MPNs). The investigators conducted a systematic review of the literature which identified several cohort and case-control studies that have investigated a wide range of potential medical, environmental and occupational risk factors. However, these studies have been limited by a wide variation in case definition and small sample sizes limiting the potential to detect modest risk differences between cases and controls. The research group propose an exploratory case-control study of 100 patients with classic MPNs and 200 controls to determine the optimal methods for roll out of this study to a multi-centred UK-based case-control study that will investigate the aetiology of MPN subtypes. The objectives of the study are to evaluate recruitment procedures, response rates and the development of a telephone administered questionnaire. The findings of this exploratory study will form the basis of a protocol for a large United Kingdom (UK)-wide case-control study of MPNs.

DETAILED DESCRIPTION:
MPNs are a group of haematopoietic malignancies resulting from a transformed haematopietic progenitor cell. They are characterised by overproduction of mature functional blood cells. MPNs were historically termed myeloproliferative disorders and have undergone numerous amendments in classification. The 2008 World Health Organisation (WHO) classifies a number of related disorders as MPNs including polycythemia vera (PV), essential thrombocythemia (ET) and primary/idiopathic myelofibrosis (PMF)2. Reported incidence rates vary from 0.02 to 2.8 per 100,000 persons3-5 but are not well characterised with half of patients asymptomatic at diagnosis6. In Northern Ireland (NI) the prevalence of ET is reported to be 18 per 100,000 persons (by correspondence, Mary McMullin). PV and ET are indolent neoplasms with better prognosis (88% and 92% 3-year survival, respectively) compared to PMF which has a 63% 3-year survival in the United States5.

The main study objectives are to:

* Develop a telephone-based questionnaire to investigate potential risk factors associated with MPNs.
* Assess the reliability and validity of the study questionnaire.
* Determine which control group to investigate by investigating:

  * Response rates.
  * Representativeness of control groups.
* Assess recruitment procedures.
* Determine if offering reimbursement of expenses (£10 per person) encourages control participation and improved representativeness to the general population.

A case-control approach was chosen as it is the most cost-efficient method of obtaining information on the aetiology of rare diseases such as MPNs. A prospective cohort study would require participation from millions of individuals followed over a long period of time. A hospital-based approach was chosen over a population-based approach to ensure the study was more feasible and could be rolled out to a number of centres in the UK.

The disorders under investigation are:

* Polycythaemia vera
* Essential Thrombocythaemia
* Primary myelofibrosis

Initially there will be one site in Belfast, Northern Ireland and one in Southampton, England. Cases will be identified and recruited through Prof Mary Frances McMullin at the Belfast City Hospital (BCH), Belfast Health and Social Care Trust, Northern Ireland and Dr Andrew Duncombe, at the University Hospital Southampton NHS Foundation Trust (UHS), Southampton, England.

Following completion of the exploratory study it is planned that other sites across the UK will be invited to participate through the Clinical Research Network.

. CASE ASCERTAINMENT Recruitment will run over a 12 month period. It is estimated that at least 100 incident and prevalent MPN cases will be recruited from the two sites during this time frame; 50 from Belfast, NI and 50 from Southampton, England. The targeted distribution of cases projected as feasible is 40 PV, 40 ET and 20 PMF cases. Fewer PMF cases are expected as the incidence is lower than PV and ET. Both incident and prevalent cases will be recruited in the exploratory case-control study and the distribution of time since diagnosis evaluated. One of the main limitations of including prevalent cases is that risk factors may differ in those who survive for a long period after diagnosis compared to those who die soon after diagnosis. Since PV and ET have low mortality rates it is expected that this will not impact the evaluation of the aetiology of these conditions to a large extent. However for PMF, which has a higher mortality rate than PV or ET, cases will be recruited as close to diagnosis as possible.

Eligible cases will be identified by the two lead clinicians Prof McMullin (Belfast) and Dr Duncombe (Southampton) during attendance at their routine clinics. Prof McMullin and Dr Duncombe will ensure that potential cases meet the study inclusion criteria (section 2.5) and provide detailed information on the categorisation of the case (PV, ET, PMF), which diagnostic criteria have been met and the clinical history of the patient.

Patients will be invited to participate in the study by letter from their lead clinician with an information sheet. Non-respondents will be randomised to either receive a reminder letter or a telephone contact from their health care team.

The choice of control group is an important consideration in any case-control study. Controls recruited from the general population through General Practitioners, population registers, neighbourhood controls or random digit dialling are ideal at identifying a representative sample of the population from which the case population was identified. However, these groups often have low response rates and selection bias is inferably encountered. Other control groups such as friend, family or hospital controls have much higher response rates but the factors associated with friendship, family or being in hospital may mean that these groups are less representative of the general population. For the purposes of this study two control groups will be recruited; GP controls and non-blood relatives (including spouses) or friend controls. The study will investigate response rates, differences in study characteristics between control groups and generalisability to the population using population-based statistics.

2.8.1 GP Controls Within each study site 5 GPs, reflective of the geographic distribution of MPN cases, will be approached to facilitate the identification and recruitment of controls and for performing phlebotomy. Each practice will be offered £200 for participation in the study.

2.8.1.1 Northern Ireland Control Recruitment in Northern Ireland will be conducted with the help of the Northern Ireland Clinical Research Network (Primary Care) (NICRN (PC)) who work in partnership with GP practices to provide support, guidance and facilitate research. The NICRN nurses who work with practices hold a Confidentiality Agreement and honorary contract with the practice. Practices are supplied with a study file, which is kept in a secure location at the practice and contains the study protocol and all relevant study information including the completed Research Governance form and contact details of researchers and NICRN (PC) staff.

With prior arrangement and agreement with the practice partners the research nurse will make an appointment with the practice manager (PM) who will either facilitate practice staff to conduct a computer search to randomly select potential controls or supply the nurse with their own unique user name and password to do so. The search will be conducted using the practice computer system's inbuilt randomisation programme, based on a numbered list of age and gender-matched patients (approximating 2 per MPN case, calculated on the basis of an attrition rate of 40-50%). The GP will be asked to confirm the eligibility of each potential control patient prior to them receiving study information from the practice.

Study information will be mailed to eligible control patients from the practice on practice headed paper and with a letter, signed by the GP, inviting them to participate. In order to track patient replies, each envelope will have a unique code number written on the front. A patient tracker form with the unique code number written beside the relevant name on the list of control patients is kept in the practice study file to track responders and non-responders for follow up purposes. No patient identifiable data will be removed from the practice at any time.

Non-respondents will be randomised to either receive a reminder letter approx two weeks after the first mail shot or to have a telephone call from practice staff using the follow-up telephone transcript.

2.8.1.2 Southampton The research nurse in Southampton will work in partnership with GP practices to provide support, guidance and facilitate research. An honorary contract and confidentiality agreement will be arranged with the practices.. This will include the nurses NMC number and copies of GCP training certificates. Practices are supplied with a study file, which is kept in a secure location at the practice and contains the study protocol and all relevant study information including the completed Research Governance form and contact details of researchers and NICRN (PC) staff.

With prior arrangement and agreement with the practice partners the research nurse will make an appointment with the practice manager (PM) who will either facilitate practice staff to conduct a computer search to randomly select potential controls or supply the nurse with their own unique user name and password to do so. The search will be conducted using the practice computer system's inbuilt randomisation programme, based on a numbered list of age and gender-matched patients (approximating 2 per MPN case, calculated on the basis of an attrition rate of 40-50%). The GP will be asked to confirm the eligibility of each potential control patient prior to them receiving study information from the practice.

Study information will be mailed to eligible control patients from the practice on practice headed paper and with a letter, signed by the GP, inviting them to participate. In order to track patient replies, each envelope will have a unique code number written on the front. A patient tracker form with the unique code number written beside the relevant name on the list of control patients is kept in the practice study file to track responders and non-responders for follow up purposes. No patient identifiable data will be removed from the practice at any time.

Non-respondents will be randomised to either receive a reminder letter approx two weeks after the first mail shot or to have a telephone call from practice staff using the follow-up telephone transcript.

2.8.2 Relative/Friend Controls Recruitment of 100 non-blood relative/friend controls will be undertaken by asking cases to pass on a flyer to up to 2 or 3 non-blood relatives/friends aged 18 years or older. Controls meeting the exclusion, section 2.7, will not be eligible for participation. Controls will not be individually matched to cases but must reside in the study area (Belfast or Southampton). Blood relatives will not be eligible for participation. Partners or friends MPN cases attending outpatient appointments in Belfast City Hospital or UHS will also be approached to participate in the study as study flyers will be available. A reminder to follow-up with recruitment of non-blood relatives/controls will be undertaken at the time of telephone interview with the cases. Those interested in participating in the study can contact the study team for the information sheet, consent form and other documentation by completing the tear off contact details strip on the flyer and posting (in the FREEPOST envelope that will be attached to the flyer) to the study team or by telephone or e-mail.

INFORMED CONSENT All cases and controls will be contacted by letter with a patient information leaflet, a consent form, patient contact form and work/residence history calendar. A pen will be included in the envelope in addition to a MPD Voice charity information sheet and a trolley token (for 50% of cases and controls). The number of subjects who refuse to participate will be documented. Subjects who refuse to participate at telephone contact will be asked whether they are willing to answer a short questionnaire to assess the representativeness of the recruited subjects. Subjects will be given the opportunity to withdraw from the study at any time however the information provided up to that point will be retained and used within the study. Subjects will be asked for verbal consent at time of telephone interview to have the interview recorded both before and after (if agreeable) the recording device is activated.

ELIGIBILITY:
Myeloproliferative neoplasm cases

Inclusion criteria:

* Clinical diagnosis of polycythemia vera, essential thrombocythaemia or primary myelofibrosis based on the WHO diagnostic criteria.
* Aged 18 years or older.

Exclusion Criteria:

* younger than 18 years old.
* where the clinician/General Practitioner (GP) does not provide consent.
* incapable of giving informed consent.
* physically or cognitively incapable of completing the questionnaire.
* too ill to participate

General Practice Controls

Inclusion Criteria:

* Randomly selected, frequency matched to the distribution of cases by 5-year age band, geographic location (Belfast and Southampton) and gender.
* Aged 18 years or older.

Exclusion Criteria:

* younger than 18 years old.
* where the clinician/GP does not provide consent.
* incapable of giving informed consent.
* physically or cognitively incapable of completing the questionnaire.
* too ill to participate.

Relative/Friend Controls

Inclusion Criteria:

* Non-blood relative/friend of a case participating in the study.
* Aged 18 years or older.

Exclusion Criteria:

* younger than 18 years old.
* where the clinician/GP does not provide consent.
* incapable of giving informed consent.
* physically or cognitively incapable of completing the questionnaire.
* too ill to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hematology clinic Primary Care clinic Non-blood relatives/ friends of cases
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley A Anderson, PhD, Principal Investigator — Queen's University, Belfast
Locations (3):
- United Kingdom (3):
  - University Hospitals Southampton NHS Foundation Trust, Southampton, England
  - Belfast Health And Social Care Trust, Belfast, Northern Ireland
  - Queen's University Belfast, Belfast, Northern Ireland

IPD SHARING:
Plan to Share IPD: Yes
Researchers can contact the study lead (Dr Anderson) to request a data access form. Once a data access form has been completed it will be reviewed by the study team and a decision made. If sharing of data has been agreed by the study team the contracts department and legal teams will review the proposed sharing of data to ensure that it meets with international standards.
Supporting Information: Study Protocol, SAP
Time Frame: Data is available from 01/09/2018 and will be available for a period of 5 years in the first instance.
Access Criteria: * Non commercial
  * Contracts/legal team to review data transfer agreements
  * Data transfer and use policy document
  * Completion of a data access form (obtainable from Dr Anderson l.anderson@qub.ac.uk)

REFERENCES:
- [Background] Anderson LA, Duncombe AS, Hughes M, Mills ME, Wilson JC, McMullin MF. Environmental, lifestyle, and familial/ethnic factors associated with myeloproliferative neoplasms. Am J Hematol. 2012 Feb;87(2):175-82. doi: 10.1002/ajh.22212. Epub 2011 Nov 11. PMID 22076943
- [Background] James G, McMullin MF, Duncombe AS, Clarke M, Anderson LA. The MOSAICC study: Assessing feasibility for biological sample collection in epidemiology studies and comparison of DNA yields from saliva and whole blood samples. Ann Hum Genet. 2018 Mar;82(2):114-118. doi: 10.1111/ahg.12227. Epub 2017 Oct 27. PMID 29076129
- [Result] Anderson LA, James G, Duncombe AS, Mesa R, Scherber R, Dueck AC, de Vocht F, Clarke M, McMullin MF. Myeloproliferative neoplasm patient symptom burden and quality of life: evidence of significant impairment compared to controls. Am J Hematol. 2015 Oct;90(10):864-70. doi: 10.1002/ajh.24098. Epub 2015 Sep 10. PMID 26113113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were invited to participate in the study by letter given to them at their clinic appointment by their clinician.
Groups:
- Myeloproliferative Neoplasm Case: Patients with Polycythemia vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF) will be recruited based on the WHO diagnostic criteria.
  Exclusion Criteria
  * younger than 18 years old.
  * where the clinician/General Practitioner (GP) does not provide consent.
  * incapable of giving informed consent.
  * physically or cognitively incapable of completing the questionnaire.
  * too ill to participate.
  Methodological pens: Randomisation of branded pen, non-branded pen and no pen
  Methodological compensation: Randomisation of a £10 monetary reimbursement for expenses on completion of the study
  Methodological trolley tokens: Trolley tokens to be randomly assigned to half of cases and General Practice controls.
- General Practice Control: For each MPN case one GP control will be randomly selected and frequency matched to the distribution of cases by 5-year age band, geographic location (Belfast and Southampton) and gender.
  The following patient groups will be excluded. Those:
  * younger than 18 years old.
  * where the clinician/GP does not provide consent.
  * incapable of giving informed consent.
  * physically or cognitively incapable of completing the questionnaire.
  * too ill to participate. The WHO performance evaluation scale will be used at the stage of participant identification. Only those scoring 0-3 will be considered eligible for inclusion in the study. Those scoring 3 are described as "Symptomatic >50% in bed but not bedbound".
  Methodological pens: Randomisation of branded pen, non-branded pen and no pen
  Methodological compensation: Randomisation of a £10 monetary reimbursement for expenses on completion of the study
  Methodological trolley tokens: Trolley tokens to be randomly assigned to half
- Non-blood Relative or Family Control: Recruitment of 100 non-blood relative/friend controls will be undertaken by asking cases to pass on a flyer to up to 2 or 3 non-blood relatives/friends aged 18 years or older.
  Methodological pens: Randomisation of branded pen, non-branded pen and no pen
  Methodological compensation: Randomisation of a £10 monetary reimbursement for expenses on completion of the study
Period: Overall Study
Arm/Group | Myeloproliferative Neoplasm Case | General Practice Control | Non-blood Relative or Family Control
Started | 106 | 47 | 81
Methodological Pens (number of those receiving pens) | 69 (37 branded pens ; 32 unbranded pens) | 29 (11 branded pens; 18 unbranded pens) | 54 (28 branded pens; 26 unbranded)
Methodological Trolley Token | 51 | 16 | 0
Methodological - £10 Cheque | 57 | 23 | 42
Initial Contact - Consent (Initial contact was via letter from clinician (cases), GP (GP controls) or info sheet (FF control)) | 84 | 35 | 81
Second Invite - Consent (Either telephone or letter as second means of contact) | 22 (9 from letter followup; 13 from phone) | 11 (2 from letter follow up; 9 from phone) | 0 (No contact info for FF controls so no second means of contact)
Completed | 106 | 45 | 81
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Myeloproliferative Neoplasm Case; General Practice Control: The letters inviting participants to participate in the study were randomised to contain:
  * a branded pen, an unbranded pen or no pen
  * a trolley token
  * Information in the study information leaflet that £10 compensation cheque would be provided upon completion and details in the letter that compensation would be provided vs no mention of compensation in the information booklet or invitation letter.
- Non-blood Relative Family Control: The letters inviting participants to participate in the study were randomised to contain:
  * a branded pen, an unbranded pen or no pen
  * Information in the study information leaflet that £10 compensation cheque would be provided upon completion and details in the letter that compensation would be provided vs no mention of compensation in the information booklet or invitation letter.
- Total: Total of all reporting groups
Arm/Group | Myeloproliferative Neoplasm Case | General Practice Control | Non-blood Relative Family Control | Total
Number analyzed (Participants) | 106 | 45 | 81 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 25 | 52 | 128
  >=65 years | 55 | 20 | 29 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.28 (12.50) | 62.10 (9.77) | 59.90 (13.52) | 61.87 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 21 | 57 | 142
  Male | 42 | 24 | 24 | 90
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 106 | 45 | 81 | 232

OUTCOME MEASURES:

1. Primary Outcome: Influence of Pre- and Post- Incentives on Participation Rates.
Description: * Difference in participation rates in those receiving:
  * vs. not receiving a pen at initial contact.
  * vs. not receiving a trolley token at initial contact.
  * vs. not receiving a monetary incentive at initial contact.
  * a MOSAICC pen vs. a non-branded pen following second contact.
  * vs. not receiving a trolley token following second contact.
  * a MOSAICC branded Pen +/or trolley token alone vs no non-monetary incentive following a second invite.
  * a MOSAICC branded Pen +/or trolley token alone vs no incentive following a second invite.
  * a MOSAICC branded Pen +/or trolley token alone vs pen/no pen &/or money following a second invite (branded vs unbranded incentive)
  * 0/1 of these incentives vs. receiving 2/3 incentives following a second invite.
  * Difference in proportion of patients completing study elements comparing:
  * 0/1 vs 2/3 incentives.
  * those receiving pre vs post invitation incentives.
Time Frame: average 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloproliferative Neoplasm Case | General Practice Control | Non-blood Relative or Family Control
Number analyzed (Participants) | 106 | 45 | 81
Participants
  No. of Participants who didn't receive an incentive | 4 | 6 | 15
  No. of participants who got pen - INITIAL CONTACT | 69 | 28 | 54
  No. participants got TrolleyToken- INITIAL CONTACT | 51 | 16 | 0
  No. participants got compensation -INITIAL CONTACT | 57 | 22 | 42
  No. who got Mosaicc pen- INITIAL CONTACT | 32 | 17 | 26
  No. who got Normal pen-INITIAL CONTACT | 37 | 11 | 28
  No. who got Pre-incentive (pen and/or trolley token) only- INITIAL CONTACT | 45 | 17 | 24
  No. who got compensation only- INITIAL CONTACT | 13 | 3 | 12
  No. who got pre & post incentive e.g. pen, trolley token and compensation - INITIAL CONTACT | 44 | 19 | 30
  No. of participants who got 0 or 1 incentive- INITIAL CONTACT | 46 | 22 | 51
  No of participants 2or 3 incentives(F/F controls could only receive a max of 2 incentives) - INITIAL | 60 | 23 | 30
  No who participated after the second invite | 24 | 10 | 0
  No of participants after second invite who initially received a MOSAICC pen | 3 | 4 | 0
  No of participants after second invite who initially received a Normal pen | 10 | 2 | 0
  No of participants after second invite who initially received a Trolley token | 14 | 6 | 0

ADVERSE EVENTS:
Time Frame: Not collected as no intervention administered
Description: Adverse Events were not collected/assessed
Groups:
- General Practice Control: For each MPN case one GP control will be randomly selected and frequency matched to the distribution of cases by 5-year age band, geographic location (Belfast and Southampton) and gender.
  The following patient groups will be excluded. Those:
  * younger than 18 years old.
  * where the clinician/GP does not provide consent.
  * incapable of giving informed consent.
  * physically or cognitively incapable of completing the questionnaire.
  * too ill to participate. The WHO performance evaluation scale will be used at the stage of participant identification. Only those scoring 0-3 will be considered eligible for inclusion in the study. Those scoring 3 are described as "Symptomatic >50% in bed but not bedbound".
Arm/Group | Myeloproliferative Neoplasm Case | General Practice Control | Non-blood Relative or Family Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No